

## **CONSENT FORM**

| HREC Project Number: | | HRE2018-0104 |
|---|---|---|
| Project Title: | | Evaluating the feasibility of providing a newly developed multifactorial falls prevention programme for community-dwelling patients after stroke. |
| Principal Investigator: | | Dr. Lex D. de Jong |
| Student researcher: | | N/A |
| Version Number: | | 1.1 |
| Version Date: | | 2018-03-05 |
| | I have read the Patient Information Statement and I understand what this project is about. | |
| | I have had an opportunity to ask questions and I am satisfied with the answers I have received. I believe I understand the purpose, extent and possible risks of my involvement in this project. | |
| | I understand that this project has been approved by Curtin University Human Research Ethics Committee and will be carried out in accordance with the National Statement on Ethical Conduct in Human Research (2007). | |
| | I voluntarily consent to take part in this research project. | |
| | I consent to being audio-recorded, photographed and video-recorded. | |
| | I understand I will receive a copy of the Patient Information Statement and Consent Form. | |
| | I consent to research data gathered for this study being used in future publications as long as my name and any other identifying information is removed. | |
| Participant Name | | |
| Participant Signature | | |
| Date | | |

## The Fall Monty Activity Programme Feasibility Study



<u>Declaration by researcher:</u> I have supplied an Information Letter and Consent Form to the participant who has signed above, and believe that they understand the purpose, extent and possible risks of their involvement in this project.

| Researcher Name |
|-------------------------|
| Researcher<br>Signature |
| Date |